CLINICAL TRIAL: NCT06995027
Title: Electrocardiographic and Echocardiographic Characteristics of Bachmann's Bundle Area Pacing
Brief Title: ECG and Echo Characteristics of BBAP
Acronym: BBAP-ECG/echo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBAP-ECG/echo
Record Dates: First submitted 2025-04-23; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pacing Therapy; Cardiac Pacing
Keywords: Bachmann's bundle pacing; Bradycardia; Physiological pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - BBAP and RAA pacing (Experimental): Bachmann's bundle area pacing (BBAP) and conventional pacing in the right atrial appendage during regular pacemaker implantation procedures are applied for acute electrocardiogram and echocardiogram testings. BBAP will be kept with remaining implantation procedure and followed-up at 3 months and/or 6 months.
  Interventions: Procedure: BBAP and RAA pacing

INTERVENTIONS:
Procedure: BBAP and RAA pacing — Bachmann's bundle area pacing and conventional pacing in the right atrial appendage during regular pacemaker implantation procedures are applied for acute electrocardiogram and echocardiogram testings.

SUMMARY:
This is a prospective, single-site, non-randomized, interventional study. The purpose is to collect electrocardiographic (ECG) and echocardiographic (echo) parameters and computed tomography (CT) images (optional) during Bachmann's bundle area pacing (BBAP) and conventional pacing in the right atrial appendage (RAA) to compare the differences between atrial pacing modalities and to further investigate the clinical outcomes of BBAP.

DETAILED DESCRIPTION:
Bachmann's bundle (BB) has emerged as an alternative pacing location to conventional right atrial appendage (RAA) pacing and is expected to avoid the interatrial conduction delay (IACD) and atrial dyssynchrony induced by RAA pacing. A recent study reported in patients with atrial pacing indications and baseline IACD that decreased atrial arrhythmia burden, recurrence, and de novo incidence were found in BB pacing, compared with right atrial septal pacing and RAA pacing. This study aimed to collect electrocardiographic (ECG) and echocardiographic (echo) parameters and CT images during BB area pacing (BBAP) and conventional pacing in the right atrial appendage (RAA) during regular pacemaker implantation procedures. The purpose is to compare the differences between atrial pacing modalities and to further investigate the clinical outcomes of BBAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 years old
* Patients who are willing to provide Informed Consent
* Patients who are indicated to atrial pacing, dual-chamber pacing, or cardiac resynchronization therapy
* Patients who consent to Bachmann's bundle area pacing

Exclusion Criteria:

* Patients who are indicated for cardiac implantable electronic device replacement or upgrade
* Patients with defibrillation indications
* Patients who are pregnant or have a plan for pregnancy during the study
* Patients who have medical conditions that would limit study participation
* Patients who were already enrolled in other trials which would impact his/her participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Atrial-paced ECG P-wave duration at implantation and during regular follow-ups | From implantation to regular follow-ups up to 6 months
Atrial-paced ECG P-wave amplitude at implantation and during regular follow-ups | From implantation to regular follow-ups up to 6 months
Atrial-paced P-onset to A-wave initiation time under Doppler at mitral and tricuspid valves at implantation | Perioperative

SECONDARY OUTCOMES:
LAD from echocardiographic measurements before implantation and during regular follow-ups | Baseline before implantation to regular follow-ups up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tong Ren Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu Z, Xianhao W, Hu W, Tang Y, Xu Z, Ou Z, Zhou Y, Ren Z, Shi T, Lu H. Interatrial Synchronized Pacing at the Posterosuperior Bundle: Feasibility, Mechanism, and Mid-Term Outcomes. Circ Arrhythm Electrophysiol. 2025 Dec 25:e014357. doi: 10.1161/CIRCEP.125.014357. Online ahead of print. PMID 41446938